CLINICAL TRIAL: NCT05537272
Title: A Study Evaluating the Therapeutic Efficacy of Tamsulosin and Tadalafil Compared to Placebo in the Treatment and Prevention of Urinary Disorders After Transperineal Prostate Biopsy
Brief Title: The Efficacy of Tamsulosin and Tadalafil Compared to Placebo in the Treatment and Prevention of Urinary Disorders After Transperineal Prostate Biopsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Ivo Juginovic, Doctor of Medicine (MD), Principal Investigator, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UHSplit
Record Dates: First submitted 2022-09-05; First posted 2022-09-13 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Lower Urinary Tract Symptoms; Voiding Disorders; Pain; Quality of Life
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Pain | interventions — Tadalafil; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Tadalafil (Active Comparator)
  Interventions: Drug: Tadalafil 5mg
- Tamsulosin (Active Comparator)
  Interventions: Drug: Tamsulosin Hydrochloride 400 Microgram Prolonged-Release Oral Capsule
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tadalafil 5mg — Administration of Tadalafil 5mg once daily seven days before and seven days after prostate biopsy
  Arms: Tadalafil
Drug: Tamsulosin Hydrochloride 400 Microgram Prolonged-Release Oral Capsule — Administration of Tamsulosin 0.4mg once daily seven days before and seven days after prostate biopsy
  Arms: Tamsulosin
Other: Placebo — Administration of placebo ( Vitamin C [ascorbic acid] 500mg tablet) once daily seven days before and seven days after prostate biopsy
  Other Names: Vitamin C (ascorbic acid) 500mg tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy of tamsulosin and tadalafil compared to placebo in the treatment and prevention of urinary disorders after transperineal prostate biopsy

DETAILED DESCRIPTION:
After being informed about the clinical study and all the risks, all patients will be given a written informed consent. They will be randomised in three groups: A (tadalafil),B (tamsulosin) and C (placebo) and the drug or placebo will be administrated seven days before and seven days after transperineal prostate biopsy. Thirty minutes before the biopsy, all patients will receive a prophylactic antibiotic (ceftriaxone 2g intravenously) and an analgetic ( naklofen 75mg intramuscular injection). Before the biopsy patients will do an uroflowmetry to determine the Qmax and ultrasound(US) of the urinary tract to determine residual urine. After the biopsy is performed the patient fills out the international prostate symptom score (IPSS/QoL), visual analog scale (VAS) for pain, International Index of Erectile Function (IIEF-5) and 36-Item Short Form Survey (SF-36) questionnaires. Seven days after the biopsy the patient discontinues with the therapy and makes a visit for routine control of uroflowmetry, US of the urinary tract and he previously mentioned questionnaires are filled out. After 30 days of the biopsy the patient makes a visit for regular control of the pathohistological findings, uroflowmetry and ultrasound of the urinary tract, along with filling out the questionnaires again.

ELIGIBILITY:
Inclusion Criteria:

* Every patient that is a candidate for first time prostate biopsy

Exclusion Criteria:

* previous complaints of the lower urinary tract; benign prostatic hyperplasia(BPH), overactive bladder (OAB), etc.
* previous urinary retention and catheterization
* previous prostate biopsies
* patients who were treated surgically or medically for BPH
* systemic diseases including uncontrolled diabetes
* neurological diseases
* hemorrhagic diathesis
* patients on anticoagulants therapy
* patients with urinary infections

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual analog scale for pain (VAS) | Time Frame 1: right after prostate biopsy, Time Frame 2: seven days after prostate biopsy
  Visual analog scale is a simple scale that rates pain form zero to ten, where zero is rated as no pain and ten is rated as unbearable pain. The patient fills it by putting an X on the lane, where no pain, mild and moderate pain is on the left side of the line and severe, very severe and worst pain possible is on the right side of the line.
Change in International prostate symptom score ( IPSS/QoL) | Time Frame 1: right after prostate biopsy, Time Frame 2: seven days after prostate biopsy, Time frame 3: 30 days after prostate biopsy
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms.
  It is a validated, reproducible scoring system to assess disease severity and response to therapy.
  The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
  There is also a separate question regarding quality of life.

SECONDARY OUTCOMES:
Change in The short form health survey - SF-36 | Time Frame 1: right after prostate biopsy, Time Frame 2: seven days after prostate biopsy, Time frame 3: 30 days after prostate biopsy
  SF -36 measure eight dimensions of quality of life: physical functioning (10 items), role limitation due to physical problems (4 items), bodily pain (2 items), social functioning (2 items), mental health (5 items), role limitation due to emotional problems (3 items), vitality (4 items) and general health perception (5 items). Each dimension has a possible score of 0 (poor health) to 100 (excellent health)
Change in The International Index of Erectile Function (IIEF-5) Questionnaire | Time Frame 1: right after prostate biopsy, Time Frame 2: seven days after prostate biopsy, Time frame 3: 30 days after prostate biopsy
  IIEF-5 is a validated questionnaire for erectile function. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
  Based on equal misclassification rates of erectile disfunction (ED) and no ED, a cutoff score of 21 (range of scores, 5-25) discriminated best. ED was classified into five severity levels, ranging from none (22-25) through severe (5-7). Substantial agreement existed between the predicted and 'true' ED classes. These data suggest that the IIEF-5 possesses favorable properties for detecting the presence and severity of ED.

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Juginović, Principal Investigator — University Hospital Split,Department of Urology; Marijan Šitum, Study Director — University Hospital Split,Department of Urology; Sandro Glumac, Study Director — University Hospital Split, Department of Anesthesiology and Intensive Care; Mario Duvnjak, Study Chair — University Hospital Split,Department of Urology; Marin Jelavić, Study Chair — University Hospital Split,Department of Urology; Ruben Kovač, Study Chair — University Hospital Split, Department of Anesthesiology and Intensive Care
Locations (1):
- University hospital of Splity, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sefik E, Eker A, Gunlusoy B, Celik S, Bozkurt IH, Basmaci I, Polat S, Degirmenci T, Ceylan Y. The effect of alpha blocker treatment prior to prostate biopsy on voiding functions, pain scores and health-related quality-of-life outcomes: A prospective randomized trial. Prog Urol. 2020 Mar;30(4):198-204. doi: 10.1016/j.purol.2019.12.006. Epub 2020 Jan 23. PMID 31983605
- [Result] Efesoy O, Saylam B, Tek M, Bozlu M, Akbay E. Is there any priority between the alpha blockers on voiding functions after transrectal ultrasound guided prostate biopsy? Turk J Urol. 2021 Mar;47(2):137-143. doi: 10.5152/tud.2021.20509. Epub 2021 Mar 1. PMID 33819444
- [Result] Chung SJ, Jung SI, Ryu JW, Hwang EC, Kwon DD, Park K, Kim JW. The preventive effect of tamsulosin on voiding dysfunction after prostate biopsy: a prospective, open-label, observational study. Int Urol Nephrol. 2015 May;47(5):711-5. doi: 10.1007/s11255-015-0955-7. Epub 2015 Mar 27. PMID 25812823
- [Result] Porst H, Oelke M, Goldfischer ER, Cox D, Watts S, Dey D, Viktrup L. Efficacy and safety of tadalafil 5 mg once daily for lower urinary tract symptoms suggestive of benign prostatic hyperplasia: subgroup analyses of pooled data from 4 multinational, randomized, placebo-controlled clinical studies. Urology. 2013 Sep;82(3):667-73. doi: 10.1016/j.urology.2013.05.005. Epub 2013 Jul 19. PMID 23876588
- [Result] Dong Y, Hao L, Shi Z, Wang G, Zhang Z, Han C. Efficacy and safety of tadalafil monotherapy for lower urinary tract symptoms secondary to benign prostatic hyperplasia: a meta-analysis. Urol Int. 2013;91(1):10-8. doi: 10.1159/000351405. Epub 2013 Jun 25. PMID 23816815
- [Result] Zisman A, Leibovici D, Kleinmann J, Cooper A, Siegel Y, Lindner A. The impact of prostate biopsy on patient well-being: a prospective study of voiding impairment. J Urol. 2001 Dec;166(6):2242-6. PMID 11696744
- [Result] Bozlu M, Ulusoy E, Doruk E, Cayan S, Canpolat B, Schellhammer PF, Akbay E. Voiding impairment after prostate biopsy: does tamsulosin treatment before biopsy decrease this morbidity? Urology. 2003 Dec;62(6):1050-3. doi: 10.1016/j.urology.2003.07.006. PMID 14665353
- [Result] Murray KS, Bailey J, Zuk K, Lopez-Corona E, Thrasher JB. A prospective study of erectile function after transrectal ultrasonography-guided prostate biopsy. BJU Int. 2015 Aug;116(2):190-5. doi: 10.1111/bju.13002. Epub 2015 Mar 23. PMID 25430505